CLINICAL TRIAL: NCT06323330
Title: Music Therapy for Rehabilitation in Post-stroke Non-fluent Aphasia: the Indian Adaptation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Institute of Human Behavior and Allied Sciences (Unknown); Indian Institute of Technology, New Delhi (Unknown); Vardhman Mahavir Medical College And Safdarjung Hospital (Other)
Responsible Party: Principal Investigator, Deepti Vibha, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-1623
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Stroke Rehabilitation; Aphasia, Broca
Keywords: Post stroke non-fluent aphasia; Melodic Intonation Therapy; Indian Adaptation
MeSH Terms: conditions — Aphasia, Broca | interventions — Rehabilitation of Speech and Language Disorders

STUDY DESIGN:
Intervention Model Description: The MIT- Indian Adaptation will be tested and compared with standard speech rehabilitation in post-stroke non-fluent aphasia
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will be given the Music Therapy, the Indian language adapted module
  Interventions: Other: Speech rehabilitation
- Active comparator (Active Comparator): The active comparator arm will be given the standard speech rehabilitation.
  Interventions: Other: Speech rehabilitation

INTERVENTIONS:
Other: Speech rehabilitation — Melodic Intonation Therapy- Indian Adaptation module which will be developed in the pilot phase

SUMMARY:
The goal of this Interventional Study is to develop and test the Indian Adaptation of Melodic Intonation Therapy (MIT) for Indian patients in with post-stroke Non-Fluent Aphasia (PSNFA). The main question[s] it aims to answer are: • To develop the MIT Indian Adaptation tool and check its feasibility • To compare the MIT with standard speech rehabilitation in patient with PSNFA. Participants will undergo Speech Rehabilitation according to the developed module and the standard treatment will be given in the comparator arm. The speech recovery at 12 weeks will be compared in both treatment arms.

DETAILED DESCRIPTION:
The study will be done in two stages:

* Stage 1 (Intervention formulation): A battery for therapy will be formulated with the help of SLT in conjunction with the expert(s) in Indian music, neurologist, and physiologist. In a series of physical and online meetings, the duration, frequency, and content of the therapy programme will be formulated. The stage(s) at which NIRS will be conducted will also be decided. This will not involve any patient recruitment and should be finished in three months.
* Stage 2 (Feasibility phase): The feasibility run will be done in 10 eligible patients. With further adaptations depending upon the experience in the feasibility phase, the pilot phase will be conducted, in which the treatment arms will be randomized.
* Stage 2 (Pilot phase): Assuming standard error of measurement for participants with aphasia as 4.33 points with a 5-point difference considered clinically meaningful for the Western Aphasia Battery (WAB), and considering that no such prior study is there, 30 patients in intervention and control arm would be initially taken. Therefore, the total sample size 10+30+30=70 patients.

  * The randomization will be done in 1:1 ratio, via a computer-generated random number sequence which will be in a sealed opaque envelope. The allocation will be concealed, and the treatment arm will be revealed after the patient has been screened and has consented for the study.
  * The outcome assessment will be by a blinded assessor, who will be a co-investigator in the study.

ELIGIBILITY:
Inclusion Criteria:

All of the following

1. Age ≥18 years of age
2. Stroke with non-fluent aphasia, within one year of ictus
3. Imaging evidence suggestive of ischemic or hemorrhagic stroke of dominant hemisphere
4. Patient is alert and able to follow simple commands (should not have global aphasia)
5. Motivated caregiver
6. Informed and signed consent

Exclusion Criteria:

Any of the following:

1. Patients with a history of a previous stroke other than the index event, which can explain the aphasia.
2. Any clinical condition (e.g., short life expectancy, coexisting disease) or other characteristics that preclude appropriate follow-up in the study (e.g., distant residence, no family support)
3. Patients participating in any therapeutic intervention clinical trials evaluating poststroke recovery
4. Use of psychotropic drugs that interfere with patient evaluation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Western Aphasia Battery Score | 8 weeks

SECONDARY OUTCOMES:
Western Aphasia Battery Score | 4 weeks
functional Near Red Spectroscopy measures | 8 weeks
modified Rankin Score | 8 weeks
Fugl Meyer Assessment Scores | 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi
  - Safdarjung Hospital, New Delhi, National Capital Territory of Delhi
  - Institute of Human Behavior and Allied Sciences, Delhi

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request to the PI